CLINICAL TRIAL: NCT00801203
Title: A Phase II/III Controlled Study to Evaluate the Effectiveness of the Induced Reflex Cough Test Plus Urodynamics to Identify Stress Urinary Incontinence in Female Subjects With a History of Stress Urinary Incontinence
Brief Title: A Study to Evaluate the Effectiveness of the Induced Reflex Cough Test Plus Urodynamics to Identify Stress Urinary Incontinence in Female Subjects With a History of Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pneumoflex Systems, LLC (Industry)
Collaborators: Ockham Development Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PNEU-01-004
Record Dates: First submitted 2008-12-01; First posted 2008-12-03 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Induced Reflex Cough Test (IRCT) followed by Voluntary Cough Test (VCT)
  Interventions: Drug: IRCT
- 2 (Experimental): Voluntary Cough Test (VCT) followed by Induced Reflex Cough Test (IRCT)
  Interventions: Drug: IRCT

INTERVENTIONS:
Drug: IRCT — Up to two administrations of the IRCT during a single cough testing session

SUMMARY:
This study is to evaluate the effectiveness of identifying stress urinary incontinence (SUI) in female subjects using the Induced Reflex Cough Test (IRCT) administered with urodynamic testing by evaluation of sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Women >25 years of age
* History of SUI (except for healthy controls)
* Healthy or stable medical problems (no change in 3 months)
* Willingness and ability to undergo all the study procedures
* Stable medications are allowed except for prescription and over-the-counter medications with anticholinergic or α-agonistic properties that can affect the bladder or urethra; these must be discontinued at least 2 weeks prior to evaluation
* Able to understand and sign the informed consent document.

Exclusion Criteria:

* Body mass index (BMI) >40
* History of severe arthritis of the hips, knees, or feet that could limit mobility during the study
* Prior treatment of any kind (surgical or pharmacologic) for incontinence at least 30 days before the cough testing session including treatment with slings, botox, interstim and all bulking agents
* Prior pelvic radiation
* Post-void residual urine >100 mL at screening
* Pelvic Organ Prolapse Quantification (POP-Q) stage >2
* Positive urine culture at screening or dip stick for >1+ leukocyte esterase on the day of the procedures
* Positive pregnancy test
* Evidence of infection with hepatitis or human immunodeficiency virus (HIV)
* Dementia
* Clinically significant changes on the electrocardiogram (ECG) in women >50 years of age or in the clinical laboratory values as determined by the investigator
* History of urge symptoms, diagnosis of interstitial cystitis, irritable bowel disease (requiring medications)
* History of neurological deficit or injury that could affect laryngeal cough reflex, for example, central nervous system related conditions such as stroke or multiple sclerosis, head and neck cancer, major laryngeal surgery
* History of neurological disorders leading to bladder abnormalities including stroke, Parkinsonism, multiple sclerosis, spinal cord surgery or spinal cord injury
* Active hemorrhoids or history of recent (within 1 year) rectal surgery
* Previous major pelvic or abdominal surgery (within 6 months)
* Tobacco smokers and non-smokers who have >15 pack-year history or frequent (>2 times per week) marijuana smoking
* Active sexually transmitted disease or genital herpes outbreak or symptomatic pelvic inflammatory disease
* Pessary in place

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity to identify SUI in women with a history of SUI and specificity to not identify SUI in healthy women without a history of SUI | Study Day 1

SECONDARY OUTCOMES:
Positive predictive value (PPV) and negative predictive value (NPV) of the IRCT administered with urodynamic testing | Study Day 1
Urodynamic parameters after IRCT and VCT in normal healthy women and women with a history of SUI | Study Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Addington, D.O., Study Director — Pneumoflex Systems, LLC
Locations (10):
- United States (10):
  - Clinical Physiology Associates, Inc, Cape Coral, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Regional Urology, LLC, Shreveport, Louisiana
  - Accumed Research Associates, Garden City, New York
  - University Urology Associates, Manhattan, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates of South Texas, McAllen, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah